CLINICAL TRIAL: NCT07303504
Title: Preparation for Sports Retirement: Protocol for a Psychoeducational Program in a Randomized Controlled Trial
Brief Title: Preparation for Sports Retirement: Study Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Sara Jiménez García-Tizón, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USAL sports retirement
Record Dates: First submitted 2025-12-10; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Sport Retirement; Psychoeducation; Retirement; Adaptation; Psychosocial Factors; Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The work of sequencing, randomisation, recruitment and allocation of the trial sample will be carried out by research staff who are not involved in the assessments or interventions of each group, thus avoiding any potential bias in the trial.
  Participants will also be blinded and will not know which group they have been allocated to and therefore which intervention they will receive. In order to minimise any contamination between groups, the assessment process will be carried out by external research staff who will perform the measurements and who have been previously trained and educated to avoid subjective bias in the process, as they will be unaware of the intervention group to which they have been assigned, thus masking the blinded assessment by third parties in the clinical trial. In addition, the researchers responsible for the statistical analysis of the trial will be blinded in order to increase the rigour of the trial process and thus the scientific quality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Programme (Active Comparator): Why: Participants will receive instructions and recommendations to facilitate a positive and healthy transition following retirement from elite sport. This minimally active intervention focuses on general guidelines for maintaining an active lifestyle and adapting to post-sport life, ensuring that the control group receives basic informational support without the structured psychoeducational sessions of the experimental group, which allows for an adequate comparison of effects. What (materials): Instructions and recommendations dossier for the program. What (procedures): Participants will be provided with a dossier containing instructions and recommendations to support the transition to sports retirement. Who will carry out the interventions: A qualified professional with experience in retirement processes will carry out the intervention. The team rotates among three professionals (psychologists specializing in retirement adjustment and a lawyer for legal aspects).
  Interventions: Behavioral: Education Programme
- Psychoeducational Programme (Experimental): Why: The program aims to facilitate a positive and healthy transition from elite sport to retirement. Its objectives include improving Quality of Life, Life Satisfaction, Psychological Flexibility, Perceived Social Support, Health, Self-Efficacy, and Self-Regulation, while simultaneously mitigating stereotypes associated with aging and the end of the sports career. What (materials): All sessions will require materials such as: projector, computer, screen, presentation of content, stationery, chairs, tables and self-recording of home tasks. What (procedures): The program combines structured education with psychoeducational activities to: Understand the retirement process and its expectations; analyze the psychosocial impact of retirement; promote physical and mental health; provide training in financial planning and benefits management; support adaptation to role changes and foster social participation; facilitate the definition and monitoring of personal goals.
  Interventions: Behavioral: Psychoeducational Programme

INTERVENTIONS:
Behavioral: Psychoeducational Programme — The program aims to facilitate a positive and healthy transition from elite sport to retirement. Its objectives include improving Quality of Life, Life Satisfaction, Psychological Flexibility, Perceived Social Support, Health, Self-Efficacy, and Self-Regulation, while simultaneously mitigating stereotypes associated with aging and the end of the sports career.
  Arms: Psychoeducational Programme
Behavioral: Education Programme — Participants will receive instructions and recommendations to facilitate a positive and healthy transition following retirement from elite sport. This minimally active intervention focuses on general guidelines for maintaining an active lifestyle and adapting to post-sport life, ensuring that the control group receives basic informational support without the structured psychoeducational sessions of the experimental group, which allows for an adequate comparison of effects.
  Arms: Education Programme

SUMMARY:
Background: This article presents the protocol for a randomised controlled trial designed to develop and evaluate a psychoeducational intervention aimed at preparing high-performance athletes for the challenges and opportunities presented by the transition to retirement from sport. The protocol was developed through a literature review and consultations with experts in sports psychology and career transition.

Methods: The study will be conducted at the Faculty of Psychology of the University of Salamanca (Spain). High-performance athletes aged 30 or older who are close to retirement or who have retired in the last five years will be recruited. Participants will be randomly assigned to two groups: the intervention group, which will undergo a psychoeducational programme consisting of 12 sessions over 3 months; and the control group, which will receive a minimum educational programme of one session. All participants will complete initial and final assessments, as well as a 3-month follow-up, collecting sociodemographic data and applying various psychological, social and health assessment instruments.

Discussion: This protocol describes a comprehensive psychoeducational intervention aimed at improving quality of life and attitudes towards retirement from sport, increasing life satisfaction, psychological flexibility, perceived social support, general health, self-efficacy and self-regulation, and reducing negative stereotypes associated with the end of a sporting career. The evidence generated will guide future interventions, policies, and educational programmes to promote a healthy, active, and satisfying transition to the post-sport stage.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they are within the critical transition period, defined as:

Five years prior to sports retirement, when the first signs of preparation and emotional anticipation begin.

Five years after retirement, the stage in which identity, psychological, and professional adaptation processes are consolidated.

This interval reflects the progressive nature of adaptation to sports retirement.

Exclusion Criteria:

* Athletes presenting any of the following conditions will be excluded from the study:

Significant literacy difficulties or relevant deficits in linguistic comprehension that prevent adequate participation in the psychoeducational sessions or the completion of assessment instruments.

Severe unstabilized medical or psychological conditions that may interfere with the normal development of the program (e.g., untreated severe depressive episodes, limiting neurological disorders).

Failure to meet the inclusion criteria, specifically not being within the five-year period prior to or after sports retirement or failing to verify high-performance sports experience.

Refusal to sign the informed consent or lack of availability to regularly attend the program sessions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Measure - Brief Version (WHOQOL-BREF) | Baseline; up to 24 weeks; 3 months follow up
  Quality of life. The range of scores is from 26 to 100 points. The higher the score, the better the quality of life.

SECONDARY OUTCOMES:
Retirement Attitudes Scale (EAJ) | Baseline; up to 24 weeks; 3 months follow up
  Attitudes towards retirement. The range of scores is from 20 to 140 points. The final scores indicate more negative attitudes the higher the value obtained
Satisfaction With Life Scale (SWLS) | Baseline; up to 24 weeks; 3 months follow up
  Satisfaction with life. The range of scores is from 5 to 25 points. A higher score indicates that the person is generally satisfied with his/her life.
Questionnaire of Stereotypes towards Old Age (CENVE) | Baseline; up to 24 weeks; 3 months follow up
  Stereotypes about ageing. The range of score is from 5 to 20 points. High scores indicate a high degree of belief in negative stereotypes of ageing.
The acceptance and action questionnaire-II (AAQ-II) | Baseline; up to 24 weeks; 3 months follow up
  Psychological inflexibility. The range of score is from 7 to 49 points. High scores indicate more psychological inflexibility.
MOS Questionnaire of Perceived Social Support (MOS) | Baseline; up to 24 weeks; 3 months follow up
  Perceived social support. The overall scores range from 20 to 100 points. The higher the score, the more social support the individual perceives.
Goldberg General Health Questionnaire (GHQ) | Baseline; up to 24 weeks; 3 months follow up
  Perceived general health. The overall scores range from 0 to 36 points. Higher scores correspond to a higher level of perceived health.
Generalised Self-Efficacy Scale (EAG) | Baseline; up to 24 weeks; 3 months follow up
  Self-efficacy. Scores range from 10 to 40 points. Higher scores indicate higher levels of self-efficacy.
Self-Regulation Scale (EAR) | Baseline; up to 24 weeks; 3 months follow up
  Self-regulation. Scores range from 7 to 35 points. Higher scores on the scale indicate a greater ability to control attention in the pursuit of goals, while lower scores may suggest difficulties in maintaining focus and attention to goals.
Athlete Retirement Questionnaire (ARQ) | Baseline; up to 24 weeks; 3 months follow up
  This measure will allow assessing the degree of planning, retirement expectations, and knowledge of available resources-all predictive factors of a more satisfactory emotional and functional adjustment (Alfermann et al., 2004). This test consists of 35 items divided into three variables: reasons for retirement (11 items), difficulties encountered during retirement (11 items), and coping strategies (13 items). The questionnaire was translated into Spanish and adapted for active athletes. It shows a Cronbach's alpha of 0.87 for the ARQ retired athletes version and 0.84 for the ARQ active athletes version. The questionnaire consists of 37 and 31 items in each of its versions respectively, with closed-ended responses.
Positive and Negative Affect Schedule (PANAS) | Baseline; up to 24 weeks; 3 months follow up
  It consists of 10 items each. Participants must indicate how much they have felt each affect on a five-point Likert scale (from 1 = not at all or very slightly to 5 = extremely) during the specified time period. The total for each scale is the summation of the scores given on the 10 items that comprise it, ranging from 10 to 50 points, where a higher score indicates a greater presence of the specific affect. The Spanish version reports high internal consistency, with a Cronbach's α of 0.87 for positive affect and 0.88 for negative affect (Vázquez et al., 2015).
Hospital Anxiety and Depression Scale (HADS) | Baseline; up to 24 weeks; 3 months follow up
  It was designed to detect anxiety and depression disorders in non-psychiatric hospital settings in patients whose symptoms were not contaminated by the symptomatology of a physical illness. It consists of 14 items grouped into two subscales with 7 items each, using a Likert-type response scale ranging from 0 to 3 points. The depression subscale is composed of items focused on anhedonia. The anxiety subscale is composed of items focused on psychic manifestations. The temporal reference for the test is the previous week. For scoring, separate scores are obtained for each of the subscales, using the following cut-off points: 0-7: normal; 8-10: probable case of anxiety or depression; 11-21: case of anxiety or depression. It possesses a Cronbach's α of 0.90 for the full scale, 0.84 for the depression subscale, and 0.85 for the anxiety subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Castilla y León, Salamanca, Salamanca 37005, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
They will be made available to researchers in the document repository "GREDOS" of the University of Salamanca, Spain.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available at the end of the study.
Access Criteria: Open access for researchers.
URL: http://gredos.usal.es/